CLINICAL TRIAL: NCT02840799
Title: Effect of KNO3 Compared to KCl on Oxygen UpTake in Heart Failure With Preserved Ejection Fraction (KNO3CK OUT HFPEF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 824290
Record Dates: First submitted 2016-06-13; First posted 2016-07-21 (Estimated); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure
Keywords: Heart Failure; Exercise Intolerance; Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — potassium nitrate; Potassium, Dietary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Potassium Nitrate (KNO3) (Experimental): Potassium nitrate (KNO3) capsules, providing 6 millimoles of inorganic nitrate per capsule, to be taken three times daily for 6 weeks.
  Interventions: Drug: Potassium Nitrate (KNO3)
- Potassium Chloride (KCl) (Placebo Comparator): Potassium Chloride (KCl) is the placebo (control drug) in this trial.
  Potassium Chloride (KCl) capsules administered at a dose of 6 millimoles (1 capsule) three times daily for 6 weeks.
  Interventions: Drug: Potassium Chloride (KCl)

INTERVENTIONS:
Drug: Potassium Nitrate (KNO3) — The effect of potassium nitrate (KNO3) supplementation on exercise capacity and peak oxygen consumption in HFpEF will be assessed.
  Arms: Potassium Nitrate (KNO3)
Drug: Potassium Chloride (KCl) — Potassium Chloride (KCl) is the matching placebo control drug in this trial.
  Arms: Potassium Chloride (KCl)

SUMMARY:
This trial seeks to assess if potassium nitrate (KNO3) therapy improves exercise capacity and oxygen uptake in heart failure patients with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
Approximately 50% of heart failure patients exhibit preserved left ventricular (LV) ejection fraction (EF), and therefore have HF with preserved EF (HFpEF). There are currently no proven effective pharmacologic interventions. Exercise intolerance with reduced aerobic capacity is the hallmark of HFpEF and greatly impairs quality of life (QOL). During exercise, blood vessels within active muscle vasodilator, increasing perfusion to the muscle bed. Nitric oxide is a chief mediator of this process. Inorganic nitrate can ultimately be converted to nitric oxide. This conversion occurs preferentially at the site of exercising muscle, allowing for vasodilation to occur, hence increasing blood flow to the working muscle. Preliminary data suggest that inorganic nitrate improves exercise tolerance in HFpEF. The investigator will aim to test this hypothesis in a larger group.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-90 years of age
2. A diagnosis of heart failure with NYHA Class II-III symptoms
3. LV ejection fraction >50% during baseline echocardiography
4. Stable medical therapy: no addition/removal/changes in antihypertensive medications, or beta-blockers in the preceding 30 days
5. Elevated filling pressures as evidenced by at least 1 of the following:

   1. Mitral E/e' ratio > 8 (either lateral or septal), with low e' velocity (septal e'<7 cm/sec or lateral e'< 10 cm/sec), in addition to one of the following:

      i Enlarged left atrium (LA volume index >34 ml/m2) ii Chronic loop diuretic use for control of symptoms iii Elevated natriuretic peptides (BNP levels >100 ng/L or NT-proBNP levels >300 ng/L)
   2. Mitral E/e' ratio > 14 (either lateral or septal)
   3. Elevated invasively-determined filling pressures previously (resting LVEDP>16 mmHg or mean pulmonary capillary wedge pressure [PCWP] > 12 mmHg; or PCWP/LVEDP≥25 mmHg with exercise)
   4. Acute heart failure decompensation requiring IV diuretics

Exclusion Criteria:

1. Supine systolic blood pressure <100 mm Hg
2. Pregnancy: Women of childbearing potential will undergo a pregnancy test during the screening visit
3. Orthostatic hypotension defined as >20 mm Hg decrease in systolic blood pressure 3-5 minutes following the transition from the supine to standing position
4. Uncontrolled atrial fibrillation, as defined by a resting heart rate>100 beats per minute
5. Hemoglobin < 10 g/dL
6. Inability/unwillingness to exercise
7. Moderate or greater left sided valvular disease (mitral regurgitation, aortic stenosis, aortic regurgitation), any degree of mitral stenosis, severe right-sided valvular disease, or presence of a prosthetic valve in the mitral position
8. Hypertrophic, infiltrative, or inflammatory cardiomyopathy
9. Clinically significant pericardial disease, as per investigator judgement.
10. Current angina
11. Acute coronary syndrome or coronary intervention within the past 2 months
12. Primary pulmonary arteriopathy
13. Clinically significant lung disease as defined by: Chronic Obstructive Pulmonary Disease meeting Stage III or greater GOLD criteria, treatment with oral steroids within the past 6 months for an exacerbation of obstructive lung disease, or the use of daytime supplemental oxygen
14. Ischemia on stress testing without either (1) subsequent revascularization, or; (2) a subsequent angiogram demonstrating the absence of clinically significant epicardial coronary artery disease, as per investigator judgement.
15. Left ventricular ejection fraction <45% in any prior echocardiogram or cardiac MRI, unless this was in the setting of uncontrolled atrial fibrillation.
16. Treatment with phosphodiesterase inhibitors that cannot be withheld
17. Treatment with organic nitrates
18. Significant liver disease impacting synthetic function or volume control (ALT/AST > 3x ULN, Albumin <3.0 g/dL)
19. eGFR < 30 mL/min/1.73m2
20. G6PD deficiency. In males of African, Asian or Mediterranean decent, this will be formally evaluated by enzyme testing prior to drug administration. A negative screening test for G6PD will be required in these subjects for inclusion in the study. If a quantitative test is being performed, a clinically significant reduction in G6PD activity (<60% of normal) will exclude subjects.
21. Methemoglobinemia - baseline methemoglobin level >5%
22. Serum K>5.0 mEq/L
23. Severe right ventricular dysfunction
24. Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the study.
25. Contraindications to MRI (except as noted below), including the presence of a pacemaker, metal implants, claustrophobia, or that have known medical conditions which can be exacerbated by stress such as anxiety or panic attacks. Inability to lie flat in the MRI scanner for 90 minutes is also an exclusion criterion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-08; Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio A Chirinos, MD, PhD, Study Chair — University of Pennsylvania; Payman Zamani, MD, Principal Investigator — University of Pennsylvania; Sanjiv Shah, MD, Principal Investigator — Northwestern University; Sujith Kuruvilla, MD, Principal Investigator — Corporal Michael J Crescenz Veterans Affairs Medical Center (VA)
Locations (3):
- United States (3):
  - Northwestern Medical Center, Evanston, Illinois
  - Corporal Michael J Crescenz Veterans Affairs Medical Center (VA), Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zamani P, Shah SJ, Cohen JB, Zhao M, Yang W, Afable JL, Caturla M, Maynard H, Pourmussa B, Demastus C, Mohanty I, Miyake MM, Adusumalli S, Margulies KB, Prenner SB, Poole DC, Wilson N, Reddy R, Townsend RR, Ischiropoulos H, Cappola TP, Chirinos JA. Potassium Nitrate in Heart Failure With Preserved Ejection Fraction: A Randomized Clinical Trial. JAMA Cardiol. 2025 Mar 1;10(3):284-289. doi: 10.1001/jamacardio.2024.4417. PMID 39693096

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following the endpoint assessment of the first phase, subjects will enter a 1-week washout period during which they will not receive any study medications.
Groups:
- Potassium Nitrate (KNO3), Then Potassium Chloride (KCl): Potassium nitrate (KNO3) capsules, provided 6 millimoles of inorganic nitrate per capsule, and was taken three times daily for 6 weeks.
  After a one week washout period, participants crossed over to take Potassium Chloride.
  Potassium Chloride (KCl) capsules was administered at a dose of 6 millimoles (1 capsule) three times daily for 6 weeks.
  Potassium Chloride (KCl): Potassium Chloride (KCl) is the matching placebo control drug in this trial.
- Potassium Chloride (KCl) Then Potassium Nitrate (KNO3): Potassium Chloride (KCl) capsules was administered at a dose of 6 millimoles (1 capsule) three times daily for 6 weeks.
  Potassium Chloride (KCl): Potassium Chloride (KCl) is the matching placebo control drug in this trial.
  Potassium Nitrate (KNO3) capsules, provided 6 millimoles of inorganic nitrate per capsule, and was taken three times daily for 6 weeks.
  After a one week washout period, participants crossed over to take Potassium Nitrate.
Period: Phase 1
Arm/Group | Potassium Nitrate (KNO3), Then Potassium Chloride (KCl) | Potassium Chloride (KCl) Then Potassium Nitrate (KNO3)
Started | 41 | 43
Completed | 36 | 40
Not Completed | 5 | 3
Not completed — Physician Decision | 1 | 3
Not completed — Withdrawal by Subject | 4 | 0
Period: Phase 2 (Crossover)
Arm/Group | Potassium Nitrate (KNO3), Then Potassium Chloride (KCl) | Potassium Chloride (KCl) Then Potassium Nitrate (KNO3)
Started (Nine participants did not cross over due to dispensing error. The subjects received the same treatment that was originally dispensed during Period 1/Phase 1.) | 41 | 35
Completed | 41 | 33
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Potassium Nitrate (KNO3) Then Potassium Chloride (KCl): Participants were randomized and first received potassium nitrate (KNO3) capsules, providing 6 millimoles of inorganic nitrate per capsule, to be taken three times daily for 6 weeks. Potassium nitrate is the active drug in this trial.
  After a washout period of 1 week, participant crossed over to receive potassium chloride (KCl), the matching placebo (control drug) in this trial. Potassium Chloride (KCl) capsules were administered at a dose of 6 millimoles (1 capsule) three times daily for 6 week.
- Experimental: Potassium Chloride (KCl) Then Potassium Nitrate (KNO3): Participants were randomized and first received potassium chloride (KCl), the matching placebo (control drug) in this trial. Potassium Chloride (KCl) capsules were administered at a dose of 6 millimoles (1 capsule) three times daily for 6 weeks.
  After a washout period of 1 week, participants cross over to receive potassium nitrate (KNO3) capsules, providing 6 millimoles of inorganic nitrate per capsule, to be taken three times daily for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Experimental: Potassium Nitrate (KNO3) Then Potassium Chloride (KCl) | Experimental: Potassium Chloride (KCl) Then Potassium Nitrate (KNO3) | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (7.55) | 67.7 (11.2) | 68.7 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 12 | 14 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 9 | 11 | 20
  White | 32 | 32 | 64
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 84
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 35.3 (7.89) | 37.1 (7.86) | 36.2 (7.88)
Current Smoker [Count of Participants; unit: Participants] — Medical history was obtained via medical chart review and participant self-reporting. Smoking status was obtained as part of their social history.
  Participants
    Yes | 0 | 0 | 0
    No | 41 | 43 | 84
Former smoker [Count of Participants; unit: Participants] — Medical history was obtained via medical chart review and participant self-reporting. Smoking status was obtained as part of their social history.
  Participants
    Yes | 24 | 14 | 38
    No | 17 | 29 | 46
Prior Acute Coronary Syndrome or Myocardial infarction [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants | 2 | 5 | 7
Prior Angina [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants | 3 | 11 | 14
Prior Arrythmia [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports. Any arrhythmia would be included in this category.
  Participants | 15 | 17 | 32
Prior significant valvular disease or valve surgery in the past [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants | 1 | 2 | 3
Hypertension [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants | 36 | 36 | 72
High Cholesterol [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants | 27 | 33 | 60
Peripheral vascular disease [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports. Peripheral vascular disease included carotid, aortic, or femoral stenosis or history of claudications.
  Participants | 3 | 2 | 5
Diabetes [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants | 17 | 21 | 38
Prior CVA/TIA [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants | 3 | 4 | 7
Prior Pulmonary embolism/DVT [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants | 4 | 2 | 6
Obstructive sleep apnea (OSA) [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants
    Obstructive sleep apnea (OSA) | 23 | 23 | 46
    CPAP Use | 17 | 17 | 34
COPD/Asthma [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants | 14 | 11 | 25
Prior CABG [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants | 2 | 3 | 5
Osteoarthritis [Count of Participants; unit: Participants] — For all participants, past medical history was obtained using chart review and participant self-reports.
  Participants | 20 | 17 | 37
NYHA Class [Count of Participants; unit: Participants] — The NYHA (New York Heart Association) classification system was used to classify participant symptoms during the baseline visit by study team.
  The following symptoms were assessed: orthopnea, paroxysmal nocturnal dyspnea, lower extremity edema, dyspnea upon exertion, and walking distance before stopping.
  With these symptoms, participants were then classified into the following NYHA classes:
  NYHA Class I = no symptoms NYHA Class II = symptoms with significant exertion NYHA Class III = symptoms with mild exertion NYHA Class IV = symptoms occur at rest
  Participants
    I | 0 | 0 | 0
    II | 33 | 25 | 58
    III | 8 | 18 | 26
    IV | 0 | 0 | 0
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — The baseline physical exam measured all vital signs.
  mmHg | 130 (16.9) | 133 (17.4) | 132 (17.1)
Diastolic Pressure [Mean (Standard Deviation); unit: mmHg] — The baseline physical exam measured all vital signs.
  mmHg | 74.7 (8.97) | 74.7 (10.2) | 74.7 (9.58)
Blood Oxygen Saturation [Mean (Standard Deviation); unit: percent (%) oxygen saturation] — The baseline physical exam measured all vital signs.
  percent (%) oxygen saturation | 97.4 (1.23) | 97.5 (1.40) | 97.5 (1.31)
6 Minute Walk Test: Total Meters Walk [Mean (Standard Deviation); unit: meters] — At the baseline visit, 6 minute walk tests were performed.
  meters | 338 (102) | 333 (94.2) | 336 (97.3)
Kansas City Cardiomyopathy Questionnaire (KCCQ) Results [Mean (Standard Deviation); unit: scores on a scale of 0-100] — KCCQ surveys were provided to participants at baseline, phase 1 visit, and phase 2 visit and scored according to KCCQ guidelines. The surveys were then scored using KCCQ guidelines, in which KCCQ scores range from 0-100, where a lower score indicates more severe symptoms/limitations and 100 indicates no symptoms.
  scores on a scale of 0-100
    Physical Limitations Score | 67.3 (16.2) | 62.0 (22.7) | 64.6 (19.9)
    Symptom Stability Score | 50.6 (14.2) | 52.3 (17.1) | 51.5 (15.7)
    Symptom Frequency Score | 69.0 (21.3) | 62.2 (24.2) | 65.5 (22.9)
    Sympton Burden Score | 69.7 (20.4) | 63.6 (21.4) | 66.6 (21)
    Total Symptom Score | 69.3 (19.6) | 62.9 (21) | 66 (20.5)
    Self-efficacy Score | 80.2 (22) | 76.5 (30.3) | 78.3 (26.5)
    Quality of Life Score | 65.0 (22.1) | 56.8 (25.8) | 60.8 (24.3)
    Social Limitation Summary Score | 57.9 (27.5) | 52.7 (23.1) | 55.3 (25.4)
    Overall Score | 64.9 (14.9) | 58.1 (18.4) | 61.4 (17)
    Clinical Summary Score | 68.3 (14) | 62.4 (18.5) | 65.3 (16.6)
Current Medications [Count of Participants; unit: Participants] — Current medications were obtained via medical chart review and participant self-reporting.
  Participants
    ACE Inhibitors | 13 | 7 | 20
    Angiotensin Receptor Blockers (ARB) | 15 | 16 | 31
    Calcium Channel Blockers (CCB) | 15 | 15 | 30
    Beta Blockers | 26 | 21 | 47
    Diuretics | 39 | 34 | 73
    Statins | 27 | 30 | 57
    Anti Arrythmia | 1 | 2 | 3
    Anti Coagulation | 2 | 0 | 2
    Anti Platelet | 28 | 29 | 57
    Insulin | 5 | 8 | 13
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] — eGFR was calculated with the 2009 CKD-EPI creatinine equation by study team. The creatinine lab results were processed during study visits.
  mL/min/1.73m^2 | 66.4 (16.6) | 70.6 (18.7) | 68.5 (17.7)
Methemeglobin [Mean (Standard Deviation); unit: Percent in blood] — During the baseline visit, participants consented to a co-oximetry blood panel, and the processing lab provided the resulting levels.
  Percent in blood | 0.729 (0.593) | 0.642 (0.379) | 0.685 (0.494)
Oxyhemoglobin [Mean (Standard Deviation); unit: Percent in blood] — During the baseline visit, participants consented to a co-oximetry blood panel, and the processing lab provided the resulting levels.
  Percent in blood | 78.5 (12.9) | 77.4 (16.7) | 77.9 (14.8)
Carboxyhemoglobin [Mean (Standard Deviation); unit: Percent in blood] — During the baseline visit, participants consented to a co-oximetry blood panel, and the processing lab provided the resulting levels.
  Percent in blood | 1.82 (0.3777) | 1.67 (0.354) | 1.75 (0.370)
O2 Count [Mean (Standard Deviation); unit: mL/dL] — During the baseline visit, participants consented to a co-oximetry blood panel, and the processing lab provided the resulting levels.
  mL/dL | 14.5 (2.64) | 15.1 (3.96) | 14.8 (3.36)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] — During the baseline visit, participants consented to a co-oximetry blood panel, and the processing lab provided the resulting levels.
  g/dL | 13.4 (1.48) | 13.6 (1.18) | 13.5 (1.33)
NT Pro-BNP [Mean (Standard Deviation); unit: pg/mL] — A sample was collected as part of visit labs and processed by our clinical laboratory for NT ProBNP
  pg/mL | 263 (332) | 213 (359) | 238 (344)
Ejection Fraction [Mean (Standard Deviation); unit: Percent total blood] — A baseline echocardiogram was performed and quantified.
  Percent total blood | 61.8 (3.92) | 61.2 (3.57) | 61.5 (3.74)
Left Atrial Volume Index [Mean (Standard Deviation); unit: mL/m^2] — A baseline echocardiogram was performed and quantified.
  mL/m^2 | 28.4 (9.45) | 26.5 (8.40) | 27.4 (8.93)
Septal E/e' Ratio [Mean (Standard Deviation); unit: Ratio] — A baseline echocardiogram was performed and quantified.
  Ratio | 14 (5.79) | 13.3 (5.39) | 13.6 (5.56)
Lateral E/e' Ratio [Mean (Standard Deviation); unit: Ratio] — A baseline echocardiogram was performed and quantified.
  Ratio | 10.1 (3.50) | 11.3 (5.34) | 10.7 (4.55)
Septal Lateral Mean E/e' Ratio [Mean (Standard Deviation); unit: Ratio] — A baseline echocardiogram was performed and quantified.
  Ratio | 11.5 (4.07) | 12.1 (4.90) | 11.8 (4.49)
White Blood Cells [Mean (Standard Deviation); unit: THO/uL] — A CBC panel was collected as part of visit labs and processed by our clinical laboratory.
  THO/uL | 6.68 (2.01) | 7.41 (1.53) | 7.06 (1.81)
Red Blood Cells [Mean (Standard Deviation); unit: MIL/uL] — A CBC panel was collected as part of visit labs and processed by our clinical laboratory.
  MIL/uL | 4.52 (0.525) | 4.56 (0.383) | 4.54 (0.455)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] — A CBC panel was collected as part of visit labs and processed by our clinical laboratory.
  g/dL | 13.2 (1.42) | 13.4 (1.15) | 13.3 (1.28)
Hematocrit [Mean (Standard Deviation); unit: Percent of blood] — A CBC panel was collected as part of visit labs and processed by our clinical laboratory.
  Percent of blood | 39.8 (4.23) | 40.5 (2.98) | 40.1 (3.63)
RDW (red blood cell distribution width) [Mean (Standard Deviation); unit: Percent red blood cells] — A CBC panel was collected as part of visit labs and processed by our clinical laboratory.
  Percent red blood cells | 14.3 (1.51) | 14.4 (1.31) | 14.3 (1.40)
MCH (mean corpuscular hemoglobin) [Mean (Standard Deviation); unit: pg] — A CBC panel was collected as part of visit labs and processed by our clinical laboratory.
  pg | 29.4 (2.74) | 19.3 (2.00) | 19.4 (2.37)
MCHC (mean corpuscular hemoglobin concentration) [Mean (Standard Deviation); unit: g/dL] — A CBC panel was collected as part of visit labs and processed by our clinical laboratory.
  g/dL | 33.1 (0.952) | 33.1 (0.930) | 33.1 (0.935)
MCV (mean corpuscular volume) [Mean (Standard Deviation); unit: fL] — A CBC panel was collected as part of visit labs and processed by our clinical laboratory.
  fL | 88.6 (7.40) | 88.8 (5.06) | 88.7 (6.26)
Platelets [Mean (Standard Deviation); unit: THO/uL] — Measure Description: A CBC panel was collected as part of visit labs and processed by our clinical laboratory.
  THO/uL | 135 (69.1) | 247 (63.7) | 241 (66.2)
Glucose [Mean (Standard Deviation); unit: mg/dL] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  mg/dL | 108 (30.9) | 112 (49.6) | 110 (41.3)
Urea Nitrogen [Mean (Standard Deviation); unit: mg/dL] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  mg/dL | 20.6 (7.76) | 10.0 (7.20) | 20.3 (7.43)
Creatinine [Mean (Standard Deviation); unit: mg/dL] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  mg/dL | 1.01 (0.230) | 1.00 (0.290) | 1.01 (0.261)
Sodium [Mean (Standard Deviation); unit: mmol/L] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  mmol/L | 139 (2.58) | 129 (2.07) | 129 (2.32)
Potassium [Mean (Standard Deviation); unit: mmol/L] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  mmol/L | 4.17 (0.435) | 4.17 (0.391) | 4.17 (0.411)
Chloride [Mean (Standard Deviation); unit: mmol/L] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  mmol/L | 101 (2.59) | 101 (3.15) | 101 (2.88)
Carbon dioxide [Mean (Standard Deviation); unit: mmol/L] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  mmol/L | 28.5 (2.84) | 28.7 (3.02) | 28.6 (2.91)
Anion gap [Mean (Standard Deviation); unit: mmol/L] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  mmol/L | 8.76 (1.39) | 8.59 (2.24) | 8.67 (1.87)
Calcium [Mean (Standard Deviation); unit: mg/dL] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  mg/dL | 9.67 (0.398) | 9.65 (0.435) | 9.66 (0.415)
Protein, total [Mean (Standard Deviation); unit: g/dL] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  g/dL | 7.13 (0.590) | 7.07 (0.501) | 7.10 (0.544)
Albumin, total [Mean (Standard Deviation); unit: g/dL] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  g/dL | 4.30 (0.291) | 4.24 (0.339) | 4.27 (0.319)
Bilirubin, total [Mean (Standard Deviation); unit: mg/dL] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  mg/dL | 0.590 (0.241) | 0.564 (0.195) | 0.577 (0.218)
Alkaline phophatase [Mean (Standard Deviation); unit: U/L] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  U/L | 78.5 (36.4) | 72.3 (19.4) | 75.3 (29.0)
AST (aspartate transferase) [Mean (Standard Deviation); unit: U/L] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  U/L | 20.5 (7.93) | 24.0 (11.5) | 22.3 (10.0)
ALT (alanine transaminase) [Mean (Standard Deviation); unit: U/L] — A CMP panel was collected as part of visit labs and processed by our clinical laboratory.
  U/L | 19.0 (8.24) | 22.2 (13.4) | 20.6 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Peak Oxygen Consumption (Vo2) Between KNO3 and KCl Phases
Description: Subjects will perform a maximal-effort peak oxygen consumption test using a supine bicycle exercise test with expired gas analysis.
Time Frame: 6 weeks after start of phase 1 (experimental drug or control); 6 weeks after start of phase 2 (experimental drug or control)
Population: As this is a crossover trial, participants received both KNO3 and KCl in different phase, and the sequence of which was dependent on a double blinded randomization. Only participants with outcome data were analyzed. The mean, SD, and t-tests were calculated based on the number of completed cases with successful crossover (N=60), but the mixed model included phase 1 data as well (N=74).
Measure: Mean (Standard Deviation); unit: L/min/kg
Groups:
- Potassium Chloride (KCl): Potassium Chloride (KCl) is the placebo (control drug) in this trial.
  Potassium Chloride (KCl) capsules administered at a dose of 6 millimoles (1 capsule) three times daily for 6 weeks.
  Potassium Chloride (KCl): Potassium Chloride (KCl) is the matching placebo control drug in this trial.
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl)
Number analyzed (Participants) | 65 | 67
L/min/kg | 10.31714 (3.851249) | 10.215172 (3.823188)
Statistical Analysis 1: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); We considered an increase in peak VO2 of ~0.6 ml/kg/min to be the minimum clinically significant change. Assuming a 90% retention rate, enrolling 84 subjects in this cross-over trial will have 80% power to detect such an effect size in the intervention induced change of our study endpoints with a two-sided α=0.05. PASS11157 was used to perform power calculations; Test type: Superiority; p = 0.6191, t-test, 2 sided — A two-sided α=0.05 was determined by the power calculation; t = -0.49979, df = 58. N=59 due to analyzing participants with complete data for Phase 1 and Phase 2 that crossovered; Mean Difference (Final Values) = -0.1309108, 95% CI 2-sided [-0.6552259 to 0.3934043], Standard Error of Mean 0.2619326 — Only participants that successfully crossed over were included in the t-test (N=59)
Statistical Analysis 2: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); The mixed model analysis provided an assessment of the treatment effect on each continuous outcome of interest while controlling for effects of other covariates such as period, sequence, and a random subject effect; Test type: Superiority; p = 0.711, Mixed Models Analysis — Assuming a 90% retention rate, enrolling 84 subjects in this cross-over trial will have 80% power to detect such an effect size in the intervention induced change of our study endpoints, with a two-sided α=0.05; Slope = 0.10, 95% CI 2-sided [-.043 to 0.62]

2. Primary Outcome: Change in Total Work Performed During a Maximal-effort Exercise Test From Phase 1 to Phase 2
Description: Subjects will perform a maximal-effort supine bicycle exercise test.
Time Frame: as for outcome 1
Population: Total work was calculated at each phase of the crossover trial. However, the analysis for the t-tests including the reported mean and standard deviation only includes cases in which Phase 1 and Phase 2 were completed.
Measure: Mean (Standard Deviation); unit: KJ
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl)
Number analyzed (Participants) | 68 | 69
KJ | 26.74341 (32.15162) | 23.76294 (29.88680)
Statistical Analysis 1: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); A two-sided α=0.05 was determined by the power calculation; Test type: Superiority; p = 0.2871, t-test, 2 sided; t = 1.0738, df = 62, p-value = 0.2871, N=63 due to analyzing participants with complete data for Phase 1 and Phase 2 that crossovered; Mean Difference (Final Values) = 2.217657, 95% CI 2-sided [-1.910612 to 6.3459261], Standard Error of Mean 2.065196
Statistical Analysis 2: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); The mixed model analysis provided an assessment of the treatment effect on each continuous outcome of interest while controlling for effects of other covariates such as period, sequence, and a random subject effect. Randomization sequence was not included in the final model due to lack of evidence for a carry over effect. Phase 1 data for participants that did not crossover due to IDS were considered for the model (N=74); Test type: Superiority; p = 0.2935, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Slope = -2.12, 95% CI 2-sided [-6.12 to 1.88]

3. Secondary Outcome: Effect of Potassium Nitrate (KNO3) on Quality of Life (QOL)
Description: QOL will be assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ). The overall summary score from the KCCQ ranges from 0-100, where higher scores indicate a better quality of life.
Time Frame: All three visits: Baseline (first) visit; 6 weeks after start of phase 1 (experimental drug or control); 6 weeks after start of phase 2 (experimental drug or control)
Population: As this is a crossover trial, participants received both KNO3 and KCl in different phases, the sequence of which was dependent on a double blinded randomization. Only participants with KCCQ results were analyzed. The mean, SD, and t-tests were calculated based on the number of completed cases with successful crossover (N=66), but the mixed model included phase 1 data as well. Baseline scores for all participants were analyzed in the mixed model as a predictive value.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Prior to randomization
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl) | Baseline
Number analyzed (Participants) | 71 | 71 | 84
score on a scale | 66.06147 (18.99883) | 62.77142 (18.95087) | 61.4335 (17.02081)
Statistical Analysis 1: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.171, t-test, 2 sided — [p-value comment as in outcome 1, analysis 2]; t=1.3844, df=65, p=0.171. N=66 due to analyzing participants with complete data for Phase 1 and Phase 2 that crossover correctly; Mean Difference (Final Values) = 2.1859922, 95% CI 2-sided [-0.9674467 to 5.3392901], Standard Error of Mean 1.578944
Statistical Analysis 2: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.113, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Slope = -2.51, 95% CI 2-sided [-5.62 to 0.61]

4. Secondary Outcome: Effect of KNO3 on the Percent Change of Systemic Vasodilatory Response to Exercise: The Change in Systemic Vascular Resistance Reserve During Exercise During a Maximal Effort Exercise Test
Description: We measured the Systematic vasodilatory response at rest and peak maximal exercise using corresponding echo parameters and blood pressures for each visit. This measure depicts the change from rest and exercise.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl)
Number analyzed (Participants) | 54 | 58
% change | -23.92288 (23.39527) | -22.13564 (24.67150)
Statistical Analysis 1: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.4905, t-test, 2 sided — [p-value comment as in outcome 1, analysis 2]; t = 0.69507, df=46, p=.4905. N=47 due to only analyzed participants that correctly crossovered; Mean Difference (Final Values) = 2.776572, 95% CI 2-sided [-5.264221 to 10.817366], Standard Error of Mean 3.99464
Statistical Analysis 2: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.796, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Slope = 1.088, 95% CI 2-sided [-7.30 to 9.48]

5. Secondary Outcome: Effect of Potassium Nitrate (KNO3) on Muscle Phosphocreatine (PCr) Recovery Kinetics Following a Standardized Plantar Flexor Exercise Protocol
Description: Muscle PCr recovery kinetics were measured using MRI and a standardized plantar flexor exercise protocol with a high resolution spatial mapping of creatine in muscle to analyze creatine chemical exchange saturation transfer and quantify the recovery kinetics of creatine levels. Exercise induces increases in the rate of O2 consumption, which upon cessation of exercise, declines towards baseline in a mono-exponential fashion. This is characterized by a time constant (τ, tau) that corresponds to the time constant of PCr recovery kinetics. Muscle PCr is a marker of oxidative capacity. This outcome measure relates to the half-time derived from linear regression, where a lower value depicts a faster PCr recovery.
Time Frame: as for outcome 1
Population: MRI was not completed throughout the duration of the study and only completed at one site (University of Pennsylvania).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl)
Number analyzed (Participants) | 15 | 15
seconds | 159.5455 (99.54442) | 219.8485 (149.41312)
Statistical Analysis 1: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.4017, t-test, 2 sided; t=-0.86929,, df=12, p=0.4017; Mean Difference (Final Values) = -38.11189, 95% CI 2-sided [-133.63637 to 57.41259], Standard Error of Mean 43.84245
Statistical Analysis 2: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.183, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Slope = 61.77, 95% CI 2-sided [-34.15 to 157.69]

6. Secondary Outcome: Effect of Potassium Nitrate (KNO3) on Left Ventricle (LV) Diastolic Function: E/e' Ratio
Description: E/e' ratio is a standard echo parameter that was measured at rest during each visit and calculated using the mitral E, septal e', and lateral e'. This index is parameter for noninvasive left ventricular diastolic function assessment, where an E/e' ratio < 8 is considered to be normal, and a ratio > 15 is considered to reflect an increase in the LV filling pressure.
Time Frame: as for outcome 3
Population: All participants were expected to undergo an echocardiogram at each visit (baseline, Phase 1, and Phase 2).
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Baseline: Prior to randomization, a baseline/screening visit was performed.
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl) | Baseline
Number analyzed (Participants) | 67 | 68 | 81
Ratio | 11.84599 (3.981865) | 11.61516 (4.265457) | 11.7999 (4.48822)
Statistical Analysis 1: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.5636, t-test, 2 sided — [p-value comment as in outcome 1, analysis 2]; t=0.58074, df=59, p=0.5636; Mean Difference (Final Values) = 0.202782, 95% CI 2-sided [-0.4959279 to 0.9014918], Standard Error of Mean 0.202782
Statistical Analysis 2: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.361, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Slope = -0.31180, 95% CI 2-sided [-0.99 to 0.37]

7. Secondary Outcome: Effect of Potassium Nitrate (KNO3) on Left Ventricle (LV) Diastolic Function: Left Atrial Volume Index
Description: Left atrial volume index is a standard echo parameter that was measured at rest during each visit and calculated the body surface area (Dubois and Dubois equation) and left atrial volume from both the two chamber and four chamber views.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl) | Baseline
Number analyzed (Participants) | 69 | 68 | 84
mL/m2 | 26.63060 (7.812431) | 27.65687 (9.931385) | 27.4408 (8.92840)
Statistical Analysis 1: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.7707, t-test, 2 sided — [p-value comment as in outcome 1, analysis 2]; t= -0.29271, df=61, p=0.7707; Mean Difference (Final Values) = -0.1532142, 95% CI 2-sided [-1.1998786 to 0.8934502], Standard Error of Mean -0.1532142
Statistical Analysis 2: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.724, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Slope = 0.18872, 95% CI 2-sided [-0.88 to 1.25]

8. Secondary Outcome: Effect of Potassium Nitrate (KNO3) on Myocardial Systolic Strain: Peak Global Systolic Myocardial Longitudinal Strain
Description: Peak global systolic myocardial longitudinal strain was evaluated with resting echocardiograms at each visit. Strain was analyzed at the four chamber, two chamber, and three chamber views of the left ventricle and averaged.
Time Frame: as for outcome 3
Population: All participants underwent an echocardiogram at each visit; however, participants in which these echo measures could not be reliably quantified were excluded.
Measure: Mean (Standard Deviation); unit: % (change in length)
Groups:
- Baseline: Prior to randomization/first visit
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl) | Baseline
Number analyzed (Participants) | 61 | 61 | 69
% (change in length) | 18.04317 (2.812165) | 17.273221 (3.003472) | 17.7164 (2.289224)
Statistical Analysis 1: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.1680825, t-test, 2 sided — [p-value comment as in outcome 1, analysis 2]; t=1.3983, df=51, p=0.1681; Mean Difference (Final Values) = 0.3262821, 95% CI 2-sided [-0.1421806 to 0.7947447], Standard Error of Mean 0.2333465
Statistical Analysis 2: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.0930, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Slope = -0.4082, 95% CI 2-sided [-0.88 to 0.07]

9. Secondary Outcome: Effect of Potassium Nitrate (KNO3) on Late Systolic Wall Stress as Assessed by the Arts Formula Using Echocardiographic and Tonometry Recordings
Description: Late systolic wall stress is assessed via comprehensive aortic pressure-flow relations, using arterial tonometry and Doppler echocardiography. Myocardial wall stress was calculated with the following formula =: Stress = P / [1/3 In (1 + VW/VLV)], where ln is the natural logarithm, P is aortic pressure obtained with arterial tonometry, VW is the volume of the LV wall obtained with echocardiography and VLV is the cavity volume obtained with echocardiography
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: dynes·cm-2·s
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl) | Baseline
Number analyzed (Participants) | 55 | 57 | 70
dynes·cm-2·s | 32.36347 (7.464010) | 34.31358 (7.837627) | 33.95494 (7.746475)
Statistical Analysis 1: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.07984, t-test, 2 sided — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = -2.116437, 95% CI 2-sided [-4.4966754 to 0.2638017], Standard Error of Mean 1.176768 — t = -1.7985, df=39, p=0.07984
Statistical Analysis 2: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.135, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Slope = 1.68, 95% CI 2-sided [-0.54 to 3.90]

10. Secondary Outcome: Effect of Potassium Nitrate (KNO3) on Arterial Wave Reflections as Assessed by Wave Separation Analysis Using Tonometry and Doppler Flow Data
Description: Arterial Wave reflections were assessed via wave separation analysis, using arterial tonometry and Doppler echocardiography.
  The pulse wave generated by the left ventricle travels forward in arteries and is partially reflected at sites of impedance mismatch (i.e., bifurcations, points of change in arterial size or wall stiffness, predominantly in middle-sized conduit arteries). Wave reflections travel back to the heart, merging into a discrete reflected wave and arrive while the LV is still ejecting blood in mid-to-late systole. Wave reflections increase the late systolic workload of the LV and profoundly impact the LV loading sequence (late relative to early systolic load).
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl) | Baseline
Number analyzed (Participants) | 55 | 57 | 70
unitless | 0.3681837 (0.08317293) | 0.372307 (0.0786807) | 0.3804 (0.07106)
Statistical Analysis 1: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.1450, t-test, 2 sided — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.0192733, 95% CI 2-sided [-0.0454871 to 0.00694040], Standard Error of Mean 0.01295984
Statistical Analysis 2: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.3047, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Slope = 0.01324, 95% CI 2-sided [-0.01 to 0.04]

11. Secondary Outcome: Effect of Potassium Nitrate (KNO3) on Augmentation Index
Description: Aortic augmentation index was assessed via comprehensive aortic pressure-flow relations, using arterial tonometry and Doppler echocardiography. It is an indirect measure of arterial stiffness, where a higher value would indicate greater arterial stiffness risk.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Index
Groups:
- Baseline: Prior to randomization/Visit 1
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl) | Baseline
Number analyzed (Participants) | 55 | 57 | 70
Index | 122.6139 (25.40388) | 122.5160 (28.58736) | 126.3574 (26.08744)
Statistical Analysis 1: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.44, t-test, 2 sided — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = -3.506681, 95% CI 2-sided [-12.598617 to 5.585256], Standard Error of Mean 4.494971
Statistical Analysis 2: Comparison: Potassium Nitrate (KNO3) vs Potassium Chloride (KCl); Test type: Superiority; p = 0.39911, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Slope = 3.39106, 95% CI 2-sided [-4.66 to 11.44]

12. Secondary Outcome: Effect of Potassium Nitrate (KNO3) on Muscle Blood Flow During Exercise: Muscle Blood Flow During Exercise, Measured With Arterial MRI Spin Labeling During a Standardized Plantar Flexion Exercise Test
Description: MRI studies will be performed at rest and immediately after a standardized plantar flexion exercise. Arterial spin labeling using the flow-sensitive alternating inversion recovery (FAIR) technique will be used to image muscle perfusion with high temporal resolution.
Time Frame: as for outcome 1
Population: Analysis could not be performed as the MRI studies were not able to extract this measure.
Arm/Group | Potassium Nitrate (KNO3), Then Potassium Chloride (KCl) | Potassium Chloride (KCl) Then Potassium Nitrate (KNO3)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Effect of Potassium Nitrate (KNO3) on Myocardial Systolic Strain: Peak Global Systolic Myocardial Circumferential Strain
Time Frame: as for outcome 3
Population: Peak Global Systolic Myocardial Circumferential Strain was not analyzed in the echocardiogram as this measure was not quantified at all during the study; instead, other strain measurements were evaluated alternatively that are considered to be more reliable.
Arm/Group | Potassium Nitrate (KNO3), Then Potassium Chloride (KCl) | Potassium Chloride (KCl) Then Potassium Nitrate (KNO3) | Baseline
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant starting on their baseline visit to 6 weeks per intervention with 1 week wash-out between, up to 13 weeks
Description: Total number at risk for baseline column is total number of participants at risk during the baseline visit including participants who screen failed (screen fail participants still attended a baseline visit). These events happened prior to randomization.
  Total number at risk for either KCl or KNO3 refers to the total number of participants randomized to medication or placebo respectively at risk for an AE.
Groups:
- Baseline Visit: At the baseline visit, patients were not on IP, but participants were monitored and consented in the study.
  All participants were at risk during their baseline visit, even the screen fails.
  Events include events that occurred in participants who were not randomized as well as those who were randomized.
Arm/Group | Potassium Nitrate (KNO3) | Potassium Chloride (KCl) | Baseline Visit
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/74 | 0/84
Serious Adverse Events (participants affected / at risk) | 1/77 | 1/74 | 1/84
Other Adverse Events (participants affected / at risk) | 43/77 | 45/74 | 61/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Potassium Nitrate (KNO3) (N=77) | Potassium Chloride (KCl) (N=74) | Baseline Visit (N=84)
abnormal sensation of swallowing (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
aches in the joints (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
acute exacerbation of bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
belching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
bilateral knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
calves aching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
creatinine increase (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0)
fever (Immune system disorders) | 0 (0) | 0 (0) | 0 (0)
flu (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
gassiness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
headache (General disorders) | 0 (0) | 0 (0) | 0 (0)
hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
hypoglycemic episode (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0)
increased stomach acid (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
nasal discharge (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0)
o2 desaturation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
oral thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
positive orthostat (General disorders) | 0 (0) | 0 (0) | 0 (0)
rapid heart beat (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
restlessness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
shortness of breath during the peak exercise test (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
stomach ache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
thigh cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
fatigue during the peak exercise test (General disorders) | 0 (0) | 0 (0) | 0 (0)
other (General disorders) | 0 (0) | 1 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Potassium Nitrate (KNO3) (N=77) | Potassium Chloride (KCl) (N=74) | Baseline Visit (N=84)
abnormal sensation of swallowing (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
aches in the joints (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
acute exacerbation of bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
belching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
bilateral knee pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
calves aching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
chest pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
creatinine increase (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (3) | 3 (3) | 3 (4)
dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
fatigue (General disorders) | 11 (12) | 4 (6) | 6 (6)
fever (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
flu (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
gassiness (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
headache (General disorders) | 8 (8) | 4 (5) | 5 (5)
hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
hypoglycemic episode (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
increased stomach acid (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
insomnia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
lightheadedness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
nasal discharge (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 6 (6) | 4 (4) | 5 (5)
nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0)
o2 desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
oral thrush (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
palpitations (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1)
positive orthostat (General disorders) | 1 (1) | 0 (0) | 0 (0)
rapid heart beat (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
restlessness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (6) | 2 (2)
shortness of breath during the peak exercise test (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
stomach ache (Gastrointestinal disorders) | 15 (18) | 7 (8) | 7 (7)
swelling (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 1 (1)
thigh cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
fatigue during the peak exercise test (General disorders) | 2 (2) | 3 (3) | 0 (0)
other (General disorders) | 16 (29) | 17 (22) | 12 (19)

LIMITATIONS AND CAVEATS:
Due to dispensing errors, nine participants didn't crossover. Overall study power was maintained. MRI completion varied across sites, leading to the discontinuation of this study component. MRI endpoints have a smaller N; interpret results cautiously. Myocardial circumferential strain wasn't quantified. Instead, longitudinal LV function, crucial for LV relaxation and filling, was quantified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT02840799/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT02840799/ICF_001.pdf